CLINICAL TRIAL: NCT06527716
Title: Exploring the Effectiveness of Applying Digital Multimedia Materials Combined With Practical Courses in Educating Clinical Nurses on Prevention of Pressure Injuries
Brief Title: Digital Multimedia in Clinical Nurse Education for Pressure Injury Prevention Via LINE@
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asia University (Other)
Responsible Party: Principal Investigator, Wen-Yi Chao, assistant professor, Asia University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AsiaU
Record Dates: First submitted 2024-07-23; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Pressure Injury
Keywords: Pressure Injury; Nurse; Knowledge,; Attitude; Self-Efficacy
MeSH Terms: conditions — Pressure Ulcer; Behavior

STUDY DESIGN:
Intervention Model Description: Control Group and Experimental Group
Who Masked: Participant
Masking Description: Participants will be aware that the teaching pertains to the prevention of pressure injuries, but they will not be informed about the specifics of the research methodology or the group assignments within the study. They will only know that this teaching is part of the in-service education program planned by the research site for that year.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional media (No Intervention): A PDF link to the pressure injury prevention course will be placed on the Nursing Information System (NIS) login interface, allowing nurses to view or download it at their convenience. A digital learning platform is also provided for downloading the self-study course materials.
- Digital multimedia combined with practical courses (Experimental): Join LINE@, which provides multimedia teaching materials and clinical scenario-based learning on a digital platform. The course includes basic knowledge learning, quizzes, and unit reviews, accessible anytime and anywhere. The digital platform continuously prompts pressure injury-related care questions and key points to stimulate learning motivation, encouraging discussion and brainstorming in the platform's discussion area.
  Interventions: Other: Teaching Strategy

INTERVENTIONS:
Other: Teaching Strategy — Experimental group:
  Get involved in the LINE digital media course learning platform.
  1. LINE digital media course study period:
     Research subjects need to complete the aforementioned three pre-measurement forms before they can join the LINE digital media course. In this lesson plan design, at the end of a single class, there will be a summary of the key points of the class; after the end of a single class, there will be 5 to 10 questions accompanying the class. When the research subjects have finished answering, Regardless of whether the answer is correct or not, the system will display "Problem Solution Analysis". The study time for this stage is 1 month.
  2. WorkShop Learning
  Control group:
  Intervention in regular education course learning platform. The above-mentioned digital media courses will be placed on the educational platform of the college for research subjects to watch and learn.
  Arms: Digital multimedia combined with practical courses

SUMMARY:
The goal of this clinical trial is to integrate past indicators affecting the effectiveness of pressure injury care education among nurses and to explore the learning outcomes of nurses through different educational interventions. The main questions it aims to answer are:

What are the outcomes of nurses' knowledge, attitudes, and self-efficacy in preventing pressure injuries after receiving education through traditional media? What are the outcomes of nurses' knowledge, attitudes, and self-efficacy in preventing pressure injuries after receiving education through digital multimedia combined with practical courses? What is the satisfaction level of nurses with pressure injury prevention education after receiving education through traditional media or digital multimedia combined with practical courses?

DETAILED DESCRIPTION:
I. Research Objectives:

To explore the effectiveness of different educational strategies on clinical nurses' prevention of pressure injuries.

II. Research Design:

A quasi-experimental design with purposive sampling, targeting clinical nurses from a regional teaching hospital. The participants are divided into a control group and an experimental group. The study focuses on pressure injury prevention, using digital media materials to present teaching content. The impact of digital media materials combined with practical courses on learning outcomes is examined. The control group will use digital media materials only, while the experimental group will use digital media materials and participate in a half-day practical course. Pre- and post-tests will be conducted for both groups before and after the course.

III. Research Subjects:

The study subjects are clinical nurses from a regional teaching hospital in central Taiwan. Inclusion criteria are: (1) full-time or part-time nursing staff registered at the research site, engaged in frontline clinical care or nursing administration, and (2) willing to participate and provide informed consent. Exclusion criteria are nursing interns. Participants who do not complete the entire training course (i.e., leave midway or terminate participation) will be excluded to avoid affecting the measurement of research outcomes.

Sample size calculation is based on G*power 3.1.7. Given that educational training has a moderate effect on nurses' knowledge and skills (Taylor-Piliae, 2008) and using Cohen's effect size analysis (Cohen, 1992), with a two-tailed test, α set at .05, power at 0.95, and effect size at 0.8, each group requires 42 samples. Considering a 40% dropout rate, 118 participants are planned, with 59 in the experimental group and 59 in the control group.

IV. Research Tools:

Digital Media Materials: Based on the 2019 international clinical practice guidelines for pressure ulcer prevention and treatment by the National Pressure Injury Advisory Panel (NPIAP), European Pressure Ulcer Advisory Panel (EPUAP), and Pan Pacific Pressure Injury Alliance (PPIAP), and the curriculum outline of the Taiwan Wound and Ostomy Care Society, four multimedia digital videos focused on pressure injury prevention are designed as the main study materials.

Demographic Data of Nurses: Including age, gender, marital status, education level, nursing rank, years of work experience, daily working hours, work unit, perceived workload, and past learning experience on pressure injuries, totaling 12 items.

Knowledge Questionnaire: Developed by Pieper and Mott in 1995 to assess healthcare workers' knowledge of pressure injury prevention. It includes questions on pressure ulcer prevention, staging, and description, with modifications to better suit healthcare settings. The final version is the 72-item Pieper-Zulkowski Pressure Ulcer Knowledge Test updated in 2021, with 31 items focused on prevention.

Attitude Questionnaire: Developed by Moore and Price in 2004 to assess nurses' attitudes toward pressure ulcer prevention. It includes 11 items rated on a Likert scale from 1 (strongly agree) to 5 (strongly disagree), with items 1, 6, 7, and 11 reverse scored. Scores range from 11 (most negative attitude) to 55 (most positive attitude).

Self-Efficacy Questionnaire: PUM-SES, published in 2019, assesses nurses' self-efficacy in managing pressure injuries. It includes 10 items across four domains: assessment, planning, supervision (two items each), and decision-making (four items). The scale uses a 5-point Likert scale, with scores ranging from 1 (cannot) to 5 (completely capable), total score from 10 to 50.

V. Research Steps:

Through verbal promotion and unit supervisor recommendation, recruit willing nursing staff to participate in the study. An information session is held to explain the research process, obtain consent, and complete pre-tests and the viewing of four multimedia digital courses on pressure injury prevention.

Control Group:

After the information session, a PDF link to the pressure injury prevention course will be placed on the Nursing Information System (NIS) login interface, allowing nurses to view or download it at their convenience. A digital learning platform is also provided for downloading the self-study course materials.

Experimental Group:

After the information session, join LINE@, which provides multimedia teaching materials and clinical scenario-based learning on a digital platform. The course includes basic knowledge learning, quizzes, and unit reviews, accessible anytime and anywhere. The digital platform continuously prompts pressure injury-related care questions and key points to stimulate learning motivation, encouraging discussion and brainstorming in the platform's discussion area.

ELIGIBILITY:
Inclusion Criteria:

1. Full-time or part-time nursing staff registered at the research site and engaged in front-line clinical care or nursing-related administrative business.
2. Those who agreed to participate in the study and provided informed consent.

Exclusion Criteria:

Nursing internship students.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Knowledge of Pressure injury | 15 minutes
  The Pressure Injury Care Cognition Scale (Pieper-Zulkowski Pressure Ulcer Knowledge Test, PZ-PUKT) was developed and tested by Pieper and Mott in 1995. The original version had 47 questions and is widely used to measure clinicians and nurses. and nursing students (Pieper & Mott, 1995). This tool is designed to assess caregivers' knowledge of pressure injuries and measures knowledge in pressure injury prevention, staging, and wound description. The question type is true or false. In addition, subjects are reminded to answer honestly. If they do not understand the question, they can choose "Unclear". Each question is scored individually. A correct answer is worth 1 point, a wrong answer or an "unclear" answer is worth 0 points; the total score is 0-31 points. The measurement process takes approximately 15 minutes.
Attitude of Pressure injury | 10 minutes
  The Attitudes to Prevent Pressure Injury Scale was derived from Moore and Price (2004) and was designed to measure nursing staff's attitudes toward preventing pressure injuries. The scale has 11 items and is scored according to a five-point Likert scale. 5 points (strongly disagree), 1 point (strongly agree) and so on. Question numbers 1, 6, 7 and 11 are reverse scored, and the points in the reverse questions range from 1 (strongly disagree) to 5 (strongly agree) and so on. The total score ranges from 11 to 55, with higher scores indicating a more positive attitude towards preventing pressure injuries.
Self-Efficacy of Pressure injury | 5 minutes
  The Pressure Injury Prevention and Management Self-Efficacy Scale is derived from Dellafiore et al. (2019). It aims to measure the self-efficacy of nurses in wound management when facing patients with pressure injuries. The scale has 10 items in total, including four Areas: There are 2 items in each of the three areas of assessment, planning and supervision, and 4 items in the decision-making area. The four areas are positively correlated. The question on the scale is: "Considering your (subject) experience working with pressure injury patients, how capable do you (subject) feel you are to face the following situations?" It is a five-point Likert scale. Scores are scored on a scale from 5 (completely in control), 1 (completely incompetent), and so on. The total score is 10-50, with higher scores indicating better self-efficacy for pressure injury prevention and management. The measurement process takes about 3-5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Hua-Shan Wu, Study Chair — Asia University

IPD SHARING:
Plan to Share IPD: No